CLINICAL TRIAL: NCT04029207
Title: The African Surgical OutcomeS-2 (ASOS-2) Trial Maternal Mortality Sub-study. A Mixed-methods Analysis of a Prospective Case-series Describing Factors Contributing to Maternal Mortality Associated With Caesarean Delivery in Africa
Brief Title: The ASOS-2 Trial Maternal Mortality Sub-study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Cape Town (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Bruce Biccard, Professor, University of Cape Town
Other Study IDs: ASOS-2 Maternal Mortality
Record Dates: First submitted 2019-06-25; First posted 2019-07-23 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Maternal Mortality; Cesarean Section; Africa
MeSH Terms: conditions — Maternal Death | interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- African Surgical OutcomeS-2 Trial: The ASOS-2 Trial is a cluster randomised trial purposively recruiting hospitals across Africa. To be eligible for inclusion a hospital must perform at least 20 cases of adult in-patient surgery with anaesthesia per week, have local ethics approval for the trial, have local hospital management approval and have established a local hospital study team. The trial excludes hospitals with lower surgical volume. The trial aims to include all consecutive adult in-patient surgical cases at participating hospitals (both elective and emergency surgery). Patients under the age of 18 and patients who have already been recruited into the trial are excluded from recruitment. Follow-up is in-hospital, censored at 30 days.
  Interventions: Procedure: Cesarean section

INTERVENTIONS:
Procedure: Cesarean section — Abdominal, operative delivery of the fetus

SUMMARY:
This sub-study is a mixed-methods analysis of a prospective case-series of maternal deaths within the African Surgical OutcomeS-2 trial cohort. The aims of the sub-study are i) to describe the contextual factors that contribute towards maternal deaths after caesarean delivery in Africa using a conceptual framework of "transport-treatment-training" and ii) to classify the maternal deaths in the ASOS-2 trial according to the WHO ICD-10 maternal mortality reporting standard. Data will be extracted from the ASOS-2 trial database. A sub-study case report form (CRF) and semi-structured telephonic interviews will be used to gather additional information from clinicians who were experienced a maternal death during the trial.

DETAILED DESCRIPTION:
This sub-study is a mixed-methods analysis of a prospective case-series of maternal deaths within the African Surgical OutcomeS-2 trial cohort. The aims of the sub-study are i) to describe the contextual factors that contribute towards maternal deaths after caesarean delivery in Africa using a conceptual framework of "transport-treatment-training" and ii) to classify the maternal deaths in the ASOS-2 trial according to the WHO ICD-10 maternal mortality reporting standard. Data will be extracted from the ASOS-2 trial database. When a maternal death is captured on the trial database, the data manager will flag the event. The hospital that registered the death will be contacted and invited to take part in the sub-study. A sub-study case report form (CRF) and semi-structured telephonic interviews will be used to gather additional information from clinicians who were experienced a maternal death during the trial.

This study uses 2 a priori frameworks for describing maternal deaths:

i) The "transport-treatment-training" framework developed by Dr Andrew Shennan (personal communication). This framework suggests that the important determinants (modifiable contextual factors) of maternal mortality can be classified as being related to transport, treatment and training factors.

* Transport refers to the manner in which the patient accesses existing care. This includes decision to seek help, modes of transportation to the hospital, and inter-facility transportation. We consider the healthcare access network in this category.
* Treatment refers to the manner in which the case was managed at the healthcare facility. It includes delays in diagnosis and decision making as well as delays between decision making and physical intervention (e.g. time from decision for caesarean delivery to time of delivery of the infant). Treatment also includes appropriateness of treatment decisions and the availability of resources needed to provide recommended treatment.
* Training refers to the availability of skilled health care providers and the need for training / upskilling of existing health care providers.

ii) The WHO application of ICD-10 codes to deaths during pregnancy, childbirth and puerperium (ICD MM) classification. Within this framework, deaths are described as having a final direct cause, an underlying cause that leads to the final cause, and contributory causes that did not directly cause death, but worsened physiological status or accelerated the underlying event.

The underlying cause of death is defined as the disease or condition that initiated the morbid chain of events leading to death or the circumstances of the accident or violence that produced a fatal injury. Underlying causes will be specified in as much detail as available. The underlying cause will be classified into one of 8 categories:

1. Hypertensive disorders in pregnancy
2. Obstetric haemorrhage
3. Pregnancy-related infection
4. Other obstetric complications
5. Unanticipated complications of management (iatrogenic)
6. Non-obstetric complications (non-obstetric disease, e.g. cardiac disease, malaria)
7. Unknown / Undetermined
8. Coincidental external causes (e.g. interpersonal violence)

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* aged 18 years and over,
* admitted to participating hospitals
* undergoing elective and non-elective caesarean delivery
* who die following their operation before leaving hospital and within 30 days after the operation.

Exclusion Criteria:

* prior participation in ASOS-2
* caesarean delivery at a hospital other than the study hospital (left censored)
* patients who are transferred to another hospital before death (right censored)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: African mothers who die during or after caesarean delivery. The primary study is a cluster randomised trial which samples hospitals across Africa purposively.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Transport: Mode of transport | On the day of hospital admission
  Nominal: walking, private transport, ambulance, public transport
Transport: Distance | On the day of hospital admission
  Continuous: distance in kilometers from patient's home to hospital
Transport: Time | On the day of hospital admission
  Continuous: time in hours from patient's home to hospital
Transport: Delay in seeking healthcare | On the day of hospital admission
  Binary: Obstetrician opinion whether there was a clinically important delay in seeking care
Transport: Delay in transport to healthcare | On the day of hospital admission
  Binary: Obstetrician opinion whether there was a clinically important delay in transport
Transport: Inter-facility delay | At time of death (death recorded in-hospital, censored at 30 days)
  Binary: Did the patient die while waiting for inter-facility transfer?
Treatment: Referral to high level of care | In-hospital censored at 30 days
  Binary: Whether or not referral to higher level of care took place
Treatment: Prophylactic uterotonic use | On day of caesarean section, at time of caesarean section
  Nominal: Oxytocin, Ergometrine, Misoprostil, Carbetocin, None
Treatment: Therapeutic uterotonic use | On day of caesarean section, at time of caesarean section
  Nominal: Oxytocin, Ergometrine, Misoprostil, Carbetocin, None
Treatment: Surgical safety checklist | On day of caesarean section, at time of caesarean section
  Binary: Whether or not a surgical safety checklist was used
Treatment: Type of anaesthetic | On day of caesarean section, at time of caesarean section
  Nominal: Regional, general with endotracheal intubation, general without endotracheal intubation.
Treatment: Airway aspiration | On day of caesarean section, at time of caesarean section
  Binary: Whether or not airway aspiration occurred
Treatment: Desaturation | On day of caesarean section, at time of caesarean section
  Binary: Whether or not desaturation below 90% occurred during management of the airway
Treatment: Spinal hypotension | On day of caesarean section, at time of caesarean section
  Binary: Whether or not spinal hypotension occured; systolic BP <= 90mmHg
Treatment: Interventions to arrest bleeding | In hospital, censored at 30 days
  Nominal: Which techniques were used? over-sowing, uterine compression suture, uterine artery ligation, uterine tourniquet, intrauterine balloon, hysterectomy, uterine artery embolisation
Treatment: Blood products | In hospital, censored at 30 days
  Nominal: Which products were given? Red blood cells, fresh frozen plasma, freeze dried plasma, cryoprecipitate, platelets, whole blood.
Treatment: Availability of medications | On day of caesarean section
  Nominal: Oxygen, Propofol, Thiopentone, Etomidate, Ketamine, Suxamethonium, Rocuronium, Nitrous Oxide, Halothane, Isoflurane, Sevoflurane, Oxytocin, Ergometrine, Syntometrine, Misoprostil, Prostaglandin F2alpha, Carbetocin, Phenylephrine, Ephedrine, Adrenalin, Noradrenalin, Morphine, Fentanyl, Pethidine, Lignocaine, Bupivacaine, Tranexamic Acid
Treatment: Availability of blood products | On day of caesarean section
  Nominal: Red blood cells, Plasma, Platelets, Cryoprecipitate
Treatment: Availability of resuscitation equipment | On day of caesarean section
  Nominal: Airway suction, endotracheal intubation equipment, mechanical ventilator, supraglottic airway devices, defibrillator,
Treatment: Availability of monitoring equipment | On day of caesarean section
  Nominal: Which monitoring equipment are available in the recovery area and the postoperative ward? O2 saturation, blood pressure, heart rate monitor, thermometer
Treatment: Recovery area | On day of caesarean section
  Binary: Is there a dedicated area where the patient is monitored during recovery from anaesthesia for caesarean section?
Treatment: Provider-patient ratio | On day of caesarean section
  Interval: Nurse-to-patient ratio in postoperative ward (during the day, during the night)
Treatment: Delay in diagnosis | On day of caesarean section
  Binary: Obstetrician opinion whether a clinical important delay in diagnosis occurred
Treatment: Delay between diagnosis and caesarean section | On day of caesarean section
  Binary: Obstetrician opinion whether a clinical important delay between diagnosis and caesarean section occurred
Treatment: Access to hospital resources | On day of caesarean section
  Nominal: Obstetrician opinion whether delayed access or lack of hospital resources contributed to the death: water supply, electricity, medications, telephone, anaesthetic equipment, surgical equipment, monitoring equipment, operating theatre, nursing or assistant, on-call senior obstetric doctor, on-call senior anaesthetic doctor, advice from referral center.
Training: Level of training | At time of caesarean section
  Nominal: Provider level of training at caesarean seciton (for anaesthesia and surgery): Specialist, specialist trainee, non-specialist doctor, non-doctor

SECONDARY OUTCOMES:
Cause of death | Maternal death is recorded in-hospital, censored at 30 days.
  WHO ICD-10 maternal mortality reporting standard

CONTACTS AND LOCATIONS:
Overall Officials: Professor Bruce M Biccard, Principal Investigator — University of Cape Town
Locations (1):
- Groote Schuur Hospital, Observatory, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Undecided
The Principle Investigator will receive requests to share individual participant data and will decide on a case by case basis.